CLINICAL TRIAL: NCT03818399
Title: Virginia Opioid Overdose Treatment InitiatVE
Acronym: VOTIVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a financial business decision by the company supporting the research study (Indivior). The decision was not due to adverse events, safety reasons, or scientific reasons, but was a business decision.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Indivior, PLC. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20015109
Record Dates: First submitted 2019-01-04; First posted 2019-01-28 (Actual); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade

STUDY DESIGN:
Intervention Model Description: The study is designed to determine effect of SUBLOCADE on repeat overdose and death compared to historical control data.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- overdose patients (Experimental): subjects that receive acute administration of SUBOXONE sublingual film in the ED followed by SUBLOCADE administration in the ED and referral to an affiliated outpatient treatment clinic, and receive monthly SUBLOCADE injections for 6 months in the context of outpatient treatment.
  Interventions: Drug: SUBLOCADE

INTERVENTIONS:
Drug: SUBLOCADE — SUBLOCADE (buprenorphine extended-release) injection is a colorless to amber sterile solution for SC injection designed to deliver buprenorphine at doses of 100 mg or 300 mg at a controlled rate over a one-month period.

SUMMARY:
This is a Phase 3b, open-label study in patients that present to the ED for an opioid OD and receive treatment with an opioid antagonist. The study is designed to determine effect of SUBLOCADE on repeat overdose and death compared to historical control data.

The study will assess subjects that receive acute administration of SUBOXONE sublingual film in the Emergency Department (ED) followed by SUBLOCADE administration in the ED and referral to an affiliated outpatient treatment clinic, compared to historical control data from electronic health records.

DETAILED DESCRIPTION:
The study will assess subjects that receive acute administration of SUBOXONE sublingual film in the Emergency Department (ED) followed by SUBLOCADE administration in the ED and referral to an affiliated outpatient treatment clinic, compared to historical control data from VCU electronic health records. The affiliated clinic will agree to see the subject on arrival at the clinic during normal clinic hours.

Patients presenting to the ED for an opioid overdose (OD) who received treatment with an opioid antagonist and are considered clinically stable and alert will be approached regarding interest in study participation. Written informed consent will only be obtained if the patient's judgement is intact as determined clinically by the investigator or a medically qualified sub-investigator or research nurse. This OD will be considered the index OD.

Subjects will be given the opportunity to participate in an optional pharmacogenetics (PGx) sub-study.

The subject will receive referral to an outpatient treatment clinic affiliated with the hospital system in which the ED resides.

Once subjects arrive at the treatment clinic, they will continue to receive SUBLOCADE for 6 months. All subjects will receive site standard psychosocial therapy at least weekly during the first 3 months of treatment, and twice monthly thereafter if clinically stable.

All subjects will complete an End of Treatment (EOT) / Early Termination (ET) visit 28 days after their last injection of SUBLOCADE. Within 3 months prior to or at the EOT visit, the investigator or a medically qualified sub-investigator will discuss the subject's available treatment options and arrange referral. All subjects will receive a safety follow-up telephone call, 30 days after their EOT/ET visit to assess AEs, SAEs, pregnancy status (if applicable) and concomitant medications. Subjects who decline to continue in medication assisted treatment (MAT) will receive monthly safety follow-up phone calls for an additional 5 months (6 months total) to assess SAEs, pregnancy status (if applicable) and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form (ICF) and have the ability to comply with the requirements and restrictions listed therein.
* Age: ≥ 18 years at time of executing the ICF.
* Currently meets DSM-5 criteria for moderate to severe opioid use disorder.
* Must have Clinical Opioid Withdrawal Scale (COWS) score of >8 to be eligible for SUBOXONE dose.
* Is clinically stable (respiratory rate [RR] ≥ 12, pulse oximetry > 95%, Glasgow Coma Scale [GCS] score of 15) and suitable for the trial in investigator or designee's judgement.
* Agrees not to take any buprenorphine products other than those administered during the current study throughout participation in the study.
* Negative urine pregnancy test for females.
* Vital signs (blood pressure, heart rate, temperature) considered within normal limits or non-clinically significant elevation, as assessed by treating physician.

Exclusion Criteria:

* Current diagnosis, other than opioid use disorder, requiring chronic opioid treatment.
* Active suicidal ideation in opinion of investigator or designee.
* Female subject that is lactating, pregnant or planning to become pregnant during their participation in the study.
* Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to provide written informed consent, signs of opioid toxicity more than 2 hours from naloxone administration or subjects with evidence of pulmonary edema.
* Known allergy or hypersensitivity to SUBOXONE.
* Any condition that, in the opinion of the investigator would interfere with interpretation of subject safety or study results.
* Currently receiving medication assisted treatment (MAT) for opioid use disorder (OUD) (e.g. methadone, buprenorphine) or received MAT as a treatment for OUD within 30 days prior to consent.
* Concurrent treatment with another investigational agent.
* Concurrent enrolment in another clinical study, or observational study that includes MAT.
* Treatment for opioid use disorder required by court order.
* Current or pending incarceration/ legal action that could affect participation or compliance in the study.
* Subjects who are unable, in the opinion of the investigator, to comply fully with the study requirements.
* Less than 48-72 hours since last use of long acting opioids (e.g., methadone), by self-report.
* Current intoxication with benzodiazepines or alcohol.
* Meet current DSM-5 diagnosis for severe Benzodiazepine or Alcohol Use Disorder, or endorse benzodiazepine or alcohol withdrawal symptoms.
* Current illicit opioid users who endorse regular use of long acting opioids (e.g. methadone).
* Total bilirubin ≥ 1.5x the upper limit of normal (ULN), alanine aminotransferase (ALT) ≥3xULN, aspartate aminotransferase (AST) ≥ 3xULN, serum creatinine > 2xULN, international normalized ratio (INR) >1.5xULN
* Patients with a history of Long QT Syndrome or an immediate family member with this condition or those taking Class lA antiarrhythmic medications (e.g., quinidine, procainamide, disopyramide) or Class Ill antiarrhythmic medications (e.g., sotalol, amiodarone, or other mediations that prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overdose Patients
Started | 19
Completed | 5
Not Completed | 14
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Overdose Patients
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Repeat OD or Opioid-related Death
Description: Repeat OD or opioid-related death will be measured from electronic medical records and state death registries
Time Frame: 6 months
Population: Because repeat OD or opioid-related death is measured from electronic medical records and state death registries, data was collected on all participants even if they did not complete the study
Measure: Count of Participants; unit: Participants
Arm/Group | Overdose Patients
Number analyzed (Participants) | 19
Participants
  Prevalence of repeat opioid-related overdose | 0
  Prevalence opioid-related death | 0

2. Secondary Outcome: Treatment Engagement
Description: Treatment engagement as measured by number of outpatient clinic visits (attendance), receipt of SUBLOCADE injections (buprenorphine treatment) at 3 and 6 months.
Time Frame: 3 and 6 months
Population: An intent to treat model was used so data from all participants, even those who did not complete, was analyzed
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Overdose Patients
Number analyzed (Participants) | 19
visits
  3 months | 8.1 (7.72)
  6 months | 13.3 (9.8)

3. Other Pre Specified Outcome: Opioid Craving
Description: Opioid craving in subjects as measured by Craving Visual Analog Scale (VAS), a 3-item scale in which individuals rate their cravings for opioids on a scale from 0 (NOT AT ALL) to 10 (EXTREMELY)
Time Frame: 6 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Illicit Opioid Use
Description: Illicit opioid use as measured by urine drug screen (UDS) results.
Time Frame: 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Genetic Predictors of Treatment Response
Description: Number of participants with mu opioid receptor polymorphisms associated with repeat overdose and death history of OD in subjects
Time Frame: 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Healthcare Resource Utilization
Description: Healthcare resource utilization (measured by number of outpatient clinic and emergency department visits, and number of inpatient admissions) as compared to the historical controls
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Treatment Effectiveness and Employment
Description: Treatment effectiveness as measured by Treatment Effectiveness Assessment (TEA)
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Medication Satisfaction
Description: measured by the Medication Satisfaction Questionnaire (MSQ)
Time Frame: 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Employment, Presentism and Absenteeism
Description: assessed by the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP)
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Overdose Patients
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overdose Patients (N=19)
Inpatient psychiatric treatment for schizoaffective disorder (Psychiatric disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overdose Patients (N=19)
Heart flutter (Cardiac disorders) | 1 (1)
Lower extremity edema (Cardiac disorders) | 1 (1)
Reduced appetite (General disorders) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1)
Inflammation at injection site (Skin and subcutaneous tissue disorders) | 1 (1)
Lip abscess (Skin and subcutaneous tissue disorders) | 1 (1)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 1 (1)
Leg muscle cramps after fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute neck strain (Musculoskeletal and connective tissue disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Injection site pain (Nervous system disorders) | 3 (5)
Acute back pain from moving (Nervous system disorders) | 1 (1)
Chronic back pain (Nervous system disorders) | 1 (1)
Chronic neck pain associated with arthritis (Nervous system disorders) | 1 (1)
Acute left knee pain with comorbid arthritis (Nervous system disorders) | 1 (1)
Sedation (General disorders) | 1 (1)
Withdrawal symptoms (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03818399/Prot_SAP_000.pdf